CLINICAL TRIAL: NCT02805322
Title: Comparison of a Novel Non-Invasive, Non-Touch Infrared Thermometer With Routine Thermometry in Routine Clinical Practice
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ARC Devices (Industry)
Collaborators: Cork University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ARC-CRFC-03
Record Dates: First submitted 2016-06-09; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Healthy; Febrile
MeSH Terms: conditions — Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Temporal Temperature Measurement (Experimental): Infrared Temporal Temperature Measurement using the ARC InstaTemp MD in three different age groups with a specified percentage reporting as febrile.
  Interventions: Device: ARC InstaTemp MD
- Tympanic and/or Sublingual Temperature (Active Comparator): Tympanic and/or Sublingual Temperature Measurement using one or both of two widely used reference clinical thermometers in three different age groups with a specified percentage reporting as febrile.
  Choice between Tympanic and/or Sublingual is determined based on standard of care in study site
  Reference Thermometer 1 - Covidien Genius 2 Tympanic Thermometer
  Reference Thermometer 2 - Welch Allen SureTemp Plus Sublingual Thermometer
  Interventions: Device: Covidien Genius 2 Tympanic Thermometer; Device: Welch Allen SureTemp Plus Sublingual Thermometer

INTERVENTIONS:
Device: ARC InstaTemp MD — Measurement of Body Temperature using an Infrared Non-Touch Thermometer - Experimental arm.
  Arms: Temporal Temperature Measurement
Device: Covidien Genius 2 Tympanic Thermometer — Measurement of Tympanic Temperature using a standard approved method - Control arm.
  Arms: Tympanic and/or Sublingual Temperature
Device: Welch Allen SureTemp Plus Sublingual Thermometer — Measurement of Sublingual Temperature using a standard approved method - Control arm.
  Arms: Tympanic and/or Sublingual Temperature

SUMMARY:
Quantify the reliability and agreement of estimated core body temperature using the InstaTemp MD™ and other widely marketed reference Thermometers

DETAILED DESCRIPTION:
This is a cross sectional Clinical Investigation in order to quantify the reliability and agreement of estimated core body temperature using emitted surface body heat measured by the InstaTemp MD™ Non-Touch thermometer when compared to other widely marketed reference Thermometers

ELIGIBILITY:
Inclusion Criteria:

1. Any age
2. Either gender
3. Attending ED, outpatients or inpatient Departments of Cork University Hospital Campus
4. Provision of informed consent or in case of minor's provision of age appropriate assent with informed consent of parent (legal guardian).

Exclusion Criteria:

1. Those who in the opinion of the researcher are too agitated, distressed or who are otherwise unable to cooperate with study procedures
2. Those who forehead cannot be fully exposed to the ambient conditions for at least 15 minutes
3. Those with signs or recent history of inflammation or infection of the forehead or at the Reference Clinical Test site
4. Subjects currently using cooling blankets or fans.
5. Subjects currently receiving treatment with thyroxine, barbiturates, antipsychotics, corticosteroids, alcoholic intoxication, documented illicit drug use or immunizations In the previous 5 days
6. Any recent hot or cold drinks prior to a sub-lingual reading (i.e. 15min before measurement)
7. Those participating in a clinical trial of an investigational medicinal product

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Mean Bias | Baseline temperature measurement using all relevant interventions
  Mean Bias (95% Levels of agreement) between ARC InstaTemp™ MD Non-Contact InfraRed Thermometry Device and (a) the Covidien Tympanic thermometer and (b) the Welch Allyn thermometer at an oral or axillary site as appropriate to subjects' age and clinical circumstance.
Reproducibility | Baseline measurement of 3 temperature reading
  Overall reproducibility of ARC InstaTemp™ MD Non-Contact InfraRed Thermometry Device.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Eustace, Prof, Principal Investigator — Cork University Hospital, Ireland
Locations (1):
- Cork University Hospital, Cork, Munster, Ireland

IPD SHARING:
Plan to Share IPD: No